CLINICAL TRIAL: NCT03994731
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Efficacy and Safety Study of Methotrexate to Increase Response Rates in Patients With Uncontrolled Gout Receiving KRYSTEXXA® (Pegloticase) (MIRROR Randomized Controlled Trial [RCT])
Brief Title: Study of KRYSTEXXA® (Pegloticase) Plus Methotrexate in Participants With Uncontrolled Gout
Acronym: MIRROR RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HZNP-KRY-202
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Gout
Keywords: gout; uncontrolled gout
MeSH Terms: conditions — Gout | interventions — Pegloticase; Methotrexate; Folic Acid; fexofenadine; Acetaminophen; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegloticase + MTX (Experimental): Following the MTX Tolerability Assessment Period (Week -6 until the Week -4 visit, in which participants take oral MTX 15 mg weekly), participants tolerating MTX are randomized to receive blinded oral MTX 15 mg weekly during the Run-in Period (from Week -4 to Day 1).
  During the Pegloticase + Immunomodulator (IMM) Period, in addition to oral 15 mg MTX, participants receive intravenous (IV) pegloticase 8 mg administered every 2 weeks (Q2W) for a total of 26 infusions from Day 1 through the Week 50 Visit.
  Per protocol, participants are also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for infusion reaction (IR) prophylaxis.
  Interventions: Biological: Pegloticase; Drug: methotrexate; Dietary Supplement: folic acid; Drug: gout flare prophylaxis regimen; Drug: fexofenadine; Drug: acetaminophen; Drug: methylprednisolone
- Pegloticase + Placebo (Placebo Comparator): Following the MTX Tolerability Assessment Period (Week -6 until the Week -4 visit, in which participants take oral MTX 15 mg weekly), participants tolerating MTX are randomized to receive blinded oral placebo for MTX weekly during the Run-in Period (from Week -4 to Day 1).
  During the Pegloticase + IMM Period, in addition to oral placebo for MTX, all participants receive IV pegloticase 8 mg administered Q2W for a total of 26 infusions from Day 1 through the Week 50 Visit.
  Per protocol, participants are also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for IR prophylaxis.
  Interventions: Biological: Pegloticase; Drug: methotrexate; Drug: placebo; Dietary Supplement: folic acid; Drug: gout flare prophylaxis regimen; Drug: fexofenadine; Drug: acetaminophen; Drug: methylprednisolone

INTERVENTIONS:
Biological: Pegloticase — IV pegloticase 8 mg Q2W
  Other Names: KRYSTEXXA®
Drug: methotrexate — Oral MTX 15 mg weekly
  Other Names: MTX
Drug: placebo — Oral placebo for MTX
  Arms: Pegloticase + Placebo
Dietary Supplement: folic acid — Folic acid 1 mg orally every day beginning at Week -6 until prior to the Week 52 Visit.
Drug: gout flare prophylaxis regimen — Prior to beginning the Pegloticase + IMM Period, participants must have been taking at least 1 protocol-standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day) for ≥ 1 week before the first dose of pegloticase and to continue flare prophylaxis per American College of Rheumatology guidelines [Khanna D et al. 2012] for the greater of 1) 6 months, 2) 3 months after achieving target serum urate (sUA < 6 mg/dL) for participants with no tophi detected on physical exam, or 3) 6 months after achieving target serum urate (sUA < 5 mg/dL) for participants with one or more tophi detected on initial physical exam that then resolved.
Drug: fexofenadine — For IR prophylaxis, fexofenadine (180 mg orally) taken the day before each infusion and on the morning of each infusion.
Drug: acetaminophen — For IR prophylaxis, acetaminophen (1000 mg orally) taken the morning of each infusion.
Drug: methylprednisolone — For IR prophylaxis, methylprednisolone (125 mg IV) given over an infusion duration between 10 - 30 minutes, immediately prior to each infusion.

SUMMARY:
The purpose of this study is to assess the potential for pegloticase with methotrexate (MTX) to increase the response rate seen with pegloticase alone, and to characterize the safety, tolerability and pharmacokinetics (PK) of the concomitant use of pegloticase with MTX, by comparing pegloticase co-administered with MTX to pegloticase co-administered with placebo for MTX in adults with uncontrolled gout.

DETAILED DESCRIPTION:
Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the study.
3. Adult men or women ≥18 years of age.
4. Uncontrolled gout, defined as meeting the following criteria:

   * Hyperuricemia during the screening period defined as sUA ≥7 mg/dL, and;
   * Failure to maintain normalization of sUA with xanthine oxidase inhibitors at the maximum medically appropriate dose, or with a contraindication to xanthine oxidase inhibitor therapy based on medical record review or subject interview, and;
   * Symptoms of gout including at least 1 of the following:

     * Presence of at least one tophus
     * Recurrent flares defined as 2 or more flares in the past 12 months prior to screening
     * Presence of chronic gouty arthritis
5. Willing to discontinue any oral urate lowering therapy for at least 7 days prior to MTX dosing at Week -6 and remain off when receiving pegloticase infusions.
6. Women of childbearing potential (including those with an onset of menopause <2 years prior to screening, non-therapy-induced amenorrhea for <12 months prior to screening, or not surgically sterile [absence of ovaries and/or uterus]) must have negative serum/urine pregnancy tests during Screening and Week -6; subjects must agree to use 2 reliable forms of contraception during the study, one of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started ≥1 full cycle prior to Week -6 (start of MTX) and continue for 30 days after the last dose of pegloticase, or at least one ovulatory cycle after the last dose of MTX or placebo for MTX (whichever is the longest duration after the last dose of pegloticase or MTX or placebo for MTX). Highly effective contraceptive methods (with a failure rate <1% per year), when used consistently and correctly, include implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or vasectomized partner.
7. Men who are not vasectomized must agree to use appropriate contraception so as to not impregnate a female partner of reproductive potential during the study, beginning with the initiation of MTX at Week -6 and continuing and for at least 3 months after the last dose of MTX or placebo for MTX.
8. Able to tolerate MTX 15 mg orally for 2 weeks (Week -6 through Week -4) prior to randomization.

Exclusion Criteria:

1. Weight >160 kg (352 pounds) at Screening.
2. Any serious acute bacterial infection, unless treated and completely resolved with antibiotics at least 2 weeks prior to the Week -6 Visit.
3. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia or chronic bronchiectasis.
4. Current or chronic treatment with systemic immunosuppressive agents such as MTX, azathioprine, or mycophenolate mofetil; prednisone ≥10 mg/day or equivalent dose of other corticosteroid on a chronic basis (3 months or longer) would also meet exclusion criteria.
5. History of any transplant surgery requiring maintenance immunosuppressive therapy.
6. Known history of hepatitis B virus surface antigen positivity or hepatitis B DNA positivity.
7. Known history of hepatitis C virus ribonucleic acid (RNA) positivity.
8. Known history of Human Immunodeficiency Virus (HIV) positivity.
9. Glucose-6-phosphate dehydrogenase deficiency (tested at the Screening Visit).
10. Chronic renal impairment defined as estimated glomerular filtration rate (eGFR) < 40 mL/min/1.73 m^2 or currently on dialysis.
11. Non-compensated congestive heart failure or hospitalization for congestive heart failure within 3 months of the Screening Visit, uncontrolled arrhythmia, treatment for acute coronary syndrome (myocardial infarction or unstable angina), or uncontrolled blood pressure (>160/100 mmHg) prior to Randomization at Week -4.
12. Pregnant, planning to become pregnant, breastfeeding, planning to impregnate female partner, or not on an effective form of birth control, as determined by the Investigator.
13. Prior treatment with pegloticase, another recombinant uricase (rasburicase), or concomitant therapy with a polyethylene glycol-conjugated drug.
14. Known allergy to pegylated products or history of anaphylactic reaction to a recombinant protein or porcine product.
15. Contraindication to MTX treatment or MTX treatment considered inappropriate.
16. Known intolerance to MTX.
17. Receipt of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to MTX administration at Week -6 or plans to take an investigational drug during the study.
18. Liver transaminase levels (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) > upper limit of normal (ULN) or albumin < the lower limit of normal (LLN) at the Screening Visit).
19. Chronic liver disease.
20. White blood cell count < 4,000/µL, hematocrit < 32 percent, or platelet count < 75,000/µL.
21. Currently receiving systemic or radiologic treatment for ongoing cancer.
22. History of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix.
23. Diagnosis of osteomyelitis.
24. Known history of hypoxanthine-guanine phosphoribosyl-transferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome.
25. Unsuitable candidate for the study, based on the opinion of the Investigator (e.g., cognitive impairment), such that participation might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or complete the study.
26. Alcohol use in excess of 3 alcoholic beverages per week.
27. A known intolerance to all protocol standard gout flare prophylaxis regimens (i.e. subject must be able to tolerate at least one: colchicine and/or non-steroidal anti inflammatory drugs and/or low dose prednisone ≤10 mg/day).
28. Current pulmonary fibrosis, bronchiectasis or interstitial pneumonitis. If deemed necessary by the Investigator, a chest X-ray may be performed during Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (60):
- United States (60):
  - University of Alabama, Birmingham, Alabama
  - Orthopedic Physicians Alaska, Anchorage, Alaska
  - Arizona Arthritis and Rheumatology Research, PLLC - Flagstaff, Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC-West, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC-East, Mesa, Arizona
  - Applied Research Center of Arkansas, Inc, Little Rock, Arkansas
  - TriWest Research Associates, El Cajon, California
  - Advanced Investigative Medicine, Inc., Hawthorne, California
  - Axis Clinical Trials, Los Angeles, California
  - ACRC Studies, Poway, California
  - ClinEdge Sierra Rheumatology, Inc., Roseville, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Providence St. John's Health Clinic, Santa Monica, California
  - Medvin Clinical Research, Tujunga, California
  - San Fernando Valley Health Institute, Van Nuys, California
  - Ventura Clinical Trials, Ventura, California
  - University of Colorado Division of Rheumatology, Aurora, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - Avail Clinical Research, DeLand, Florida
  - Prohealth Research Center, Doral, Florida
  - Omega Research Maitland, Orlando, Florida
  - DMI Research, Pinellas Park, Florida
  - Napa Research Center, Pompano Beach, Florida
  - GCP Clinical Research, Tampa, Florida
  - Florida Medical Clinic, LLC, Zephyrhills, Florida
  - St. Luke's Clinic - Rheumatology, Meridian, Idaho
  - MD Medical Research, Oxon Hill, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Infusion Associates, Grand Rapids, Michigan
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - Benefis Hospital, Great Falls, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Santa Fe Rheumatology, Santa Fe, New Mexico
  - Long Island Arthritis & Osteoporosis Care, Babylon, New York
  - Buffalo Rheumatology and Medicine, Orchard Park, New York
  - NorthEast Rheumatology/Atrium Health, Concord, North Carolina
  - NorthEast Rheumatology, Concord, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - ClinEdge PMG Research of Hickory, LLC, Hickory, North Carolina
  - ClinEdge PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Shelby Clinical Research, LLC, Shelby, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Premier Clinical/STAT Research, Dayton, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Clinical Research Source Inc., Perrysburg, Ohio
  - Premier Clinical/STAT Research - Springboro, Springboro, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - Articularis Healthcare Group, Summerville, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C. Gupta, M.D., Memphis, Tennessee
  - Diagnostic and Interventional Nephrology Of Houston, Houston, Texas
  - Research Consultants - Frostwood, Houston, Texas
  - Research Consultants - Astoria, Houston, Texas
  - Arthritis Clinic of Central Texas, San Marcos, Texas
  - Arthritis & Osteoporosis Clinic - Waco, Waco, Texas
  - Clear Lake Specialties, Webster, Texas
  - Western Washington Arthritis Clinic, Bothell, Washington
  - Arthritis Northwest, Spokane, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Botson J, Obermeyer K, LaMoreaux B, Padnick-Silver L, Verma S, Weinblatt ME, Peterson J. Quality of life and clinical gout assessments during pegloticase with and without methotrexate co-therapy: MIRROR randomized controlled trial exploratory findings. Rheumatol Adv Pract. 2024 Nov 29;8(4):rkae145. doi: 10.1093/rap/rkae145. eCollection 2024. PMID 39678124
- [Derived] Dalbeth N, Botson J, Saag K, Kumar A, Padnick-Silver L, LaMoreaux B, Becce F. Monosodium urate crystal depletion and bone erosion remodeling during pegloticase treatment in patients with uncontrolled gout: Exploratory dual-energy computed tomography findings from MIRROR RCT. Joint Bone Spine. 2024 Jul;91(4):105715. doi: 10.1016/j.jbspin.2024.105715. Epub 2024 Mar 4. PMID 38447697
- [Derived] Botson JK, Saag K, Peterson J, Parikh N, Ong S, La D, LoCicero K, Obermeyer K, Xin Y, Chamberlain J, LaMoreaux B, Verma S, Sainati S, Grewal S, Majjhoo A, Tesser JRP, Weinblatt ME. A Randomized, Placebo-Controlled Study of Methotrexate to Increase Response Rates in Patients with Uncontrolled Gout Receiving Pegloticase: Primary Efficacy and Safety Findings. Arthritis Rheumatol. 2023 Feb;75(2):293-304. doi: 10.1002/art.42335. Epub 2022 Dec 16. PMID 36099211

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 2-week MTX Tolerability Assessment Period consisting of 2 weeks oral MTX. 159 participants received MTX in this period. The 7 participants who were unable to tolerate MTX in this period or who met other exclusion criteria were not randomized, were classified as screen failures, and were not considered enrolled per protocol section 9.4.6.3.2.2. 152 randomized participants were considered enrolled in this trial.
Groups:
- Pegloticase + MTX: Participants were randomized to receive blinded oral MTX 15 mg weekly during the Run-in Period. During the Pegloticase + Immunomodulator (IMM) Period, in addition to oral MTX 15 mg, participants received intravenous (IV) pegloticase 8 mg every 2 weeks (Q2W) for a total of 26 infusions from Day 1 through the Week 50 Visit.
  Per protocol, participants were also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for infusion reaction (IR) prophylaxis.
- Pegloticase + Placebo: Participants were randomized to receive blinded oral MTX 15 mg weekly during the Run-in Period. During the Pegloticase + IMM Period, in addition to oral placebo for MTX, participants received IV pegloticase 8 mg Q2W for a total of 26 infusions from Day 1 through the Week 50 Visit.
  Per protocol, participants were also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for IR prophylaxis.
Period: Run-in Period (From Week -4 to Day 1)
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Started (Randomized) | 100 | 52
Took at Least 1 Dose of MTX or Placebo | 98 | 51
Completed | 96 | 49
Not Completed | 4 | 3
Period: Pegloticase + IMM Period
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Started | 96 | 49
Completed | 76 | 34
Not Completed | 20 | 15
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- Pegloticase + MTX: Participants were randomized to receive blinded oral MTX 15 mg weekly during the Run-in Period. During the Pegloticase + IMM Period, in addition to oral MTX 15 mg, participants received IV pegloticase 8 mg Q2W for a total of 26 infusions from Day 1 through the Week 50 Visit.
  Per protocol, participants were also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for IR prophylaxis.
- Total: Total of all reporting groups
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo | Total
Number analyzed (Participants) | 100 | 52 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.74) | 53.0 (12.12) | 54.7 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 91 | 44 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 9 | 28
  Not Hispanic or Latino | 81 | 42 | 123
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Black or African American | 16 | 6 | 22
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  White | 69 | 36 | 105
  Other, Not Specified | 3 | 2 | 5
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Serum Uric Acid (sUA) Responders (sUA < 6 mg/dL) During Month 6
Description: Responders are defined as participants achieving and maintaining sUA < 6 mg/dL for at least 80% of the time during Month 6. Month 6 includes pre- and post-infusion sUA assessments at Weeks 20 and 22, non-infusion sUA at Weeks 21 and 23, pre-infusion sUA at Week 24 and any unscheduled sUA between Week 20 and Week 24. A participant must have had ≥ 2 sUA observations from different visits in order to be eligible as a responder. Participants meeting the stopping rule (those with a pre-infusion sUA >6 mg/dL at 2 consecutive scheduled trial visits beginning with the Week 2 Visit stopped pegloticase dosing) were counted as non-responders.
Time Frame: Month 6 (Weeks 20, 21, 22, 23 and 24)
Population: Intent-to-treat (ITT) Population: all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Number analyzed (Participants) | 100 | 52
percentage of participants | 71.0 [61.1 to 79.6] | 38.5 [25.3 to 53.0]
Statistical Analysis 1: Comparison: Pegloticase + MTX vs Pegloticase + Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — The 2-sided p-value was calculated assuming the test statistic was distributed as a standard normal random variable; Stratified difference in proportions = 32.31, 95% CI 2-sided [16.3 to 48.3], Standard Error of Mean 8.157 — Stratified difference (Pegloticase+MTX - Pegloticase+Placebo) is a weighted average of the difference within each stratum. Estimates from the 2 strata (tophi presence at baseline: yes, no) were combined with Cochran-Mantel-Haenszel (CMH) weights

2. Secondary Outcome: Percentage of sUA (sUA < 6 mg/dL) Responders During Month 12
Description: Responders are defined as participants achieving and maintaining sUA <6 mg/dL for at least 80% of the time during Month 12 (Weeks 48, 50 and 52). Month 12 includes pre- and post-infusion sUA Weeks 48 and 50, pre-infusion sUA at Week 52, and any unscheduled sUA assessments done at unscheduled visits between Week 48 and 52. A participant must have had ≥ 2 sUA observations from different visits in order to be eligible as a responder. Participants meeting the stopping rule (those with a pre-infusion sUA >6 mg/dL at 2 consecutive scheduled trial visits beginning with the Week 2 Visit stopped pegloticase dosing) were counted as non-responders.
Time Frame: Month 12 (Weeks 48, 50 and 52)
Population: ITT Population: all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Number analyzed (Participants) | 100 | 52
percentage of participants | 60.0 [49.7 to 69.7] | 30.8 [18.7 to 45.1]
Statistical Analysis 1: Comparison: Pegloticase + MTX vs Pegloticase + Placebo; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — The 2-sided p-value was calculated assuming the test statistic was distributed as a standard normal random variable; response rate difference = 29.05, 95% CI 2-sided [13.2 to 44.9], Standard Error of Mean 8.084 — response rate difference (Peg+MTX - Peg+Placebo)

3. Secondary Outcome: Percentage of Participants With Complete Resolution of ≥ 1 Tophi at Week 52
Description: Percentage of participants with complete resolution of ≥ 1 tophi (using digital photography) at Week 52 in participants with tophi at baseline. Participants with resolution of ≥ 1 tophi at a visit are participants with resolution of ≥ 1 tophi at the visit (i.e. have complete response), and no progressive disease for any other tophi.
Time Frame: Baseline, Week 52
Population: ITT Population: all randomized participants with ≥ 1 tophi at baseline. Modified non-responder imputation was done for participants with missing tophi evaluation data at Week 52.
Measure: Number; unit: percentage of participants
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Number analyzed (Participants) | 52 | 29
percentage of participants | 53.8 | 31.0
Statistical Analysis 1: Comparison: Pegloticase + MTX vs Pegloticase + Placebo; Test type: Superiority; p = 0.0482, Chi-squared — The comparison of complete response between groups is performed using an unstratified chi-squared test; Difference = 22.8, 95% CI 2-sided [1.2 to 44.4] — Difference (Pegloticase+MTX - Pegloticase+Placebo)

4. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 52
Description: HAQ-DI is a self-report functional status instrument that is filled out by the participant and measures disability over the past week via 20 questions relating to 8 domains of function: dressing, grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. The HAQ-DI ranges from 0 to 3 with higher values indicating higher disability. A change from baseline value of 0 is imputed at the first post-baseline visit for any participants without post-baseline values.
Time Frame: Baseline, Week 52
Population: ITT Population: all randomized participants. Participants with an assessment at Week 52.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Number analyzed (Participants) | 76 | 34
score on a scale | -0.35 (0.049) | -0.31 (0.071)
Statistical Analysis 1: Comparison: Pegloticase + MTX vs Pegloticase + Placebo; Test type: Superiority; p = 0.6287, MMRM ANCOVA — Based on mixed models repeated measures (MMRM) analysis of covariance (ANCOVA) model including the following terms: baseline value, tophi presence (Y/N), treatment group, visit, visit-by-treatment interaction, and visit-by-baseline value interaction; Difference = -0.04, 95% CI 2-sided [-0.21 to 0.13], Standard Error of Mean 0.084 — Difference (Pegloticase+MTX - Pegloticase+Placebo)

5. Secondary Outcome: Mean Change From Baseline HAQ Pain Score at Week 52
Description: The HAQ-Pain score rates the participant's pain over the past week from 0 to 100 with 0 = no pain and 100 = severe pain. A change from baseline value of 0 is imputed at the first post-baseline visit for any participants without post-baseline values.
Time Frame: Baseline, Week 52
Population: ITT Population: all randomized participants. Participants with an assessment at Week 52.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Number analyzed (Participants) | 76 | 34
score on a scale | -31.02 (2.208) | -22.59 (3.230)
Statistical Analysis 1: Comparison: Pegloticase + MTX vs Pegloticase + Placebo; Test type: Superiority; p = 0.0272, MMRM ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference = -8.43, 95% CI 2-sided [-15.88 to -0.97], Standard Error of Mean 3.766 — Difference (Pegloticase+MTX - Pegloticase+Placebo)

6. Secondary Outcome: Mean Change From Baseline in HAQ Health Score at Week 52
Description: The HAQ health scale is a self-reported measure of overall health. Participants are asked to rate how they are doing, considering all the ways arthritis affects them, on a scale of 0 to 100, where 0 represents very well and 100 represents very poor. A change from baseline value of 0 is imputed at the first post-baseline visit for any participants without post-baseline values.
Time Frame: Baseline, Week 52
Population: ITT Population: all randomized participants. Participants with an assessment at Week 52.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pegloticase + MTX | Pegloticase + Placebo
Number analyzed (Participants) | 76 | 34
score on a scale | -28.85 (2.531) | -18.69 (3.722)
Statistical Analysis 1: Comparison: Pegloticase + MTX vs Pegloticase + Placebo; Test type: Superiority; p = 0.0222, MMRM ANCOVA — [p-value comment as in outcome 4, analysis 1]; Difference = -10.16, 95% CI 2-sided [-18.84 to -1.48], Standard Error of Mean 2.531 — Difference (Pegloticase+MTX - Pegloticase+Placebo)

ADVERSE EVENTS:
Time Frame: All Cause Mortality: from signing of informed consent up to Week 52 plus 30 days after last pegloticase infusion (±3 days). Adverse events (AEs)in the Run-in Period: Week -6 up to Day 1 (predose). AEs in the Pegloticase + IMM Period: Day 1 up to Week 52 plus 30 days after last pegloticase infusion (±3 days).
Description: The number of participants at risk is not consistent with the Participant Flow data table because the 7 participants who were not randomized after receiving MTX during the 2-week MTX Tolerability Assessment Period were not considered enrolled.
Groups:
- MTX: Methotrexate Tolerability Assessment Period: Participants received open-label oral MTX 15 mg for 2 weeks. Participants not tolerating MTX were designated as screen failures).
- Pegloticase + MTX: Run-In Period; Pegloticase + Placebo: Run-In Period: Participants were randomized to receive blinded oral MTX 15 mg weekly during the Run-in Period.
  Per protocol, participants were also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for IR prophylaxis.
- Pegloticase + MTX: Pegloticase + IMM Period: Participants were randomized to receive blinded oral MTX 15 mg weekly during the Run-in Period. During the Pegloticase + IMM Period, in addition to oral MTX 15 mg, participants received IV pegloticase 8 mg Q2W for a total of 26 infusions from Day 1 through the Week 50 Visit.
  Per protocol, participants were also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for IR prophylaxis.
- Pegloticase + Placebo: Pegloticase + IMM Period: Participants were randomized to receive blinded oral MTX 15 mg weekly during the Run-in Period. During the Pegloticase + IMM Period, in addition to oral placebo for MTX, participants received IV pegloticase 8 mg Q2W for a total of 26 infusions from Day 1 through the Week 50 Visit.
  Per protocol, participants were also required to take folic acid, at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day), and a regimen of fexofenadine, acetaminophen, and methylprednisolone for IR prophylaxis.
Arm/Group | MTX: Methotrexate Tolerability Assessment Period | Pegloticase + MTX: Run-In Period | Pegloticase + Placebo: Run-In Period | Pegloticase + MTX: Pegloticase + IMM Period | Pegloticase + Placebo: Pegloticase + IMM Period
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/98 | 0/51 | 2/96 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/159 | 1/98 | 0/51 | 13/96 | 5/49
Other Adverse Events (participants affected / at risk) | 45/159 | 28/98 | 10/51 | 71/96 | 42/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTX: Methotrexate Tolerability Assessment Period (N=159) | Pegloticase + MTX: Run-In Period (N=98) | Pegloticase + Placebo: Run-In Period (N=51) | Pegloticase + MTX: Pegloticase + IMM Period (N=96) | Pegloticase + Placebo: Pegloticase + IMM Period (N=49)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 2
Abscess Soft Tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MTX: Methotrexate Tolerability Assessment Period (N=159) | Pegloticase + MTX: Run-In Period (N=98) | Pegloticase + Placebo: Run-In Period (N=51) | Pegloticase + MTX: Pegloticase + IMM Period (N=96) | Pegloticase + Placebo: Pegloticase + IMM Period (N=49)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4
Fatigue (General disorders) | 0 | 0 | 0 | 5 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 7 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 13
Gout (Metabolism and nutrition disorders) | 45 | 28 | 10 | 64 | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 13 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT03994731/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT03994731/SAP_001.pdf